CLINICAL TRIAL: NCT02209077
Title: Repeatability and Reproducibility of Optic Nerve Head (ONH), Retinal Nerve Fiber Layer (RNFL), and Macula Parameters With the Heidelberg Spectralis OCT.
Brief Title: Spectralis OCT Repeatability and Reproducibility Study
Acronym: S-2013-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-2013-1 Study (REPRO)
Record Dates: First submitted 2013-08-12; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Experimental): OCT performed to collect data from the back of the eye
  Interventions: Device: OCT performed to collect data from the back of the eye
- Glaucoma group (Experimental): OCT performed to collect data from the back of the eye
  Interventions: Device: OCT performed to collect data from the back of the eye

INTERVENTIONS:
Device: OCT performed to collect data from the back of the eye — comparative retinal parameters with Spectralis OCT

SUMMARY:
This single-center, prospective, interventional clinical study is conducted to evaluate the repeatability and reproducibility of structural parameters of the optic nerve head, the peripapillary retinal nerve fiber layer, and the macula using the Heidelberg Spectralis OCT (Optical Coherence Tomography) device. Data obtained from healthy volunteers in this study are compared to those from a previous, larger healthy volunteer study that was conducted in the United States and Europe (S-2012-1), and data from glaucoma patients are compared to those from the healthy volunteers.

DETAILED DESCRIPTION:
The study will include approximately 15 normal subjects and approximately 15 subjects who have glaucoma of varying degree. All subjects will undergo Spectralis OCT imaging and other study procedures in one single visit. All examinations performed on the subjects are non-significant risk procedures because the medical devices are cleared for marketing in Europe and in the U.S. Total study duration is anticipated to not exceed 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject is not an employee of the eye clinic.
* Age ≥18
* Able and willing to undergo the test procedures, give consent, and to follow instructions.
* For "normal subjects": Healthy eye without prior intraocular surgery (except cataract surgery and Lasik - laser-assisted refractive surgery) and without clinically significant vitreal, retinal or choroidal diseases, diabetic retinopathy, or disease of the optic nerve.
* For "glaucoma subjects": Early to advanced glaucoma according to existing medical charts.
* Refraction between +6 and -6 diopters and astigmatism ≤ 2 diopters.
* When both eyes are eligible, one randomly selected eye will enter the study.

Exclusion Criteria:

• Insufficient quality of Spectralis OCT images (this is not determined until after Spectralis OCT examination, and is an unusual circumstance). Minimum requirements are:

* Retina completely included in image frame,
* Quality Score ≥ 20 in the stored ART mean images

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Reproducibility and repeatability of multiple parameters (measured with OCT in the back of the eye) between different studies and different subject types | one day
  This study is designed to determine optic nerve head structural values such as ONH rim thickness, RNFL thickness values, and macula structural values such as total retinal or ganglion cell layer thickness, as measured using the Spectralis device in a population of either subjects that are determined to be clinically "normal" or "glaucomatous". The expected reproducibility and repeatability are approximately 5% or less of the respective means (coefficients of variation, cov). This study shall result in a 95% confidence interval of the cov estimate not larger than ±1% when all data is pooled (normal and glaucoma cases). Statistical analysis of the measurement values will consist of the computation of mean and standard deviation in repeated examinations with the SPECTRALIS OCT in the normal and glaucomatous population.

CONTACTS AND LOCATIONS:
Overall Officials: Balwantray C Chauhan, PhD, Principal Investigator — Department of Ophthalmology and Visual Sciences, Dalhousie University, Halifax, Canada
Locations (1):
- Department of Ophthalmology and Visual Sciences, Dalhousie University, Halifax, Nova Scotia, Canada